CLINICAL TRIAL: NCT05225545
Title: Randomized Controlled Trial of Sucrosomial Iron vs. Oral Iron Sulfate for the Treatment of Iron Deficiency Anemia in Patients With Ulcerative Colitis
Brief Title: Sucrosomial Iron vs. Oral Iron Sulfate for the Treatment of Iron Deficiency Anemia in Patients With Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Pharma M SAL, Lebanon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2019-0046:
Record Dates: First submitted 2020-10-09; First posted 2022-02-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Anemia, Iron Deficiency; Ulcerative Colitis
Keywords: Sucrosomial Iron; Sideral Forte; Iron Supplementation; Iron Deficiency; Anemia; Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Anemia, Iron-Deficiency; Colitis, Ulcerative; Iron Deficiencies; Anemia; Inflammatory Bowel Diseases | interventions — sucrosomial iron; Iron

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrosomial Iron (Experimental): These patients will receive Sucrosomial Iron 30 mg + 70 mg ascorbic acid (Sideral Forte) twice daily
  Interventions: Drug: Sucrosomial Iron
- Oral Iron Therapy (Active Comparator): These patients will receive Oral Iron therapy at a dose of 195 mg twice daily for the same period of time
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Sucrosomial Iron — Experimental Arm
  Other Names: Sideral Forte
  Arms: Sucrosomial Iron
Drug: Oral Iron — Active Comparator
  Arms: Oral Iron Therapy

SUMMARY:
The aim of the study is to compare the tolerability and efficacy of Sucrosomial Iron to Oral Iron Therapy in a randomized controlled trial for the treatment of Iron Deficiency Anemia in Ulcerative Colitis patients.

DETAILED DESCRIPTION:
Ulcerative Colitis (UC) is an inflammatory bowel disease (IBD) characterized by chronic inflammation limited to the mucosal layer of the colon. Anemia is a consistent clinical feature of IBD, and is encountered in one third of patients [1] and Anemia in Ulcerative Colitis is most commonly the result of iron-deficiency due to chronic blood loss through ulcerations in the colon.

Oral Iron supplementation has been used for the treatment of Iron Deficiency anemia but may cause disease exacerbation in patients with UC [2]. Iron also can increase cancer risk [3], and is associated with many side effects such as constipation, diarrhea, nausea, vomiting, abdominal pain and hyperchromia of feces. Furthermore, studies have shown that oral iron supplementation fails to resolve anemia in 2 of 3 IBD patients. [4]

Sucrosomial iron is a new preparation of iron pyrophosphate delivered within a phospholipid membrane and coated with sucrester (sucrose esters of fatty acids). it has been shown to have better absorption and higher bioavailability while minimizing side effects in multiple patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Confirmed diagnosis of Ulcerative Colitis
* Proven Iron Deficiency Anemia (Hb < 12 for females and Hb < 13 for males AND iron saturation <20%)
* Hemoglobin level > 8g/dl

Exclusion Criteria:

* Age below 18
* Hemoglobin level < 8g/dl
* Recently hospitalized for disease flare (within 3 months)
* Hemoglobinopathies (including thalassemia)
* Isolated proctitis
* Indeterminate colitis
* Known liver or kidney disease
* Known Celiac Disease
* Extensive small bowel resection
* Use of anticoagulants or aspirin
* Known intolerance to oral iron therapy
* Uninvestigated anemia
* Pregnant or lactating women
* Known hypersensitivity to iron sulfate
* Transfusion in the past 4 weeks
* Erythropoetin within the last 8 weeks
* Rheumatoid Arthritis
* History of menometrorrhagia or frequent epistaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
Tolerability of experimental product | 12 weeks
  Tolerability will be assessed via a Treatment Tolerability Assessment Questionnaire

SECONDARY OUTCOMES:
Response to iron repletion | 12 weeks
  Hemoglobin
Compliance and adherence | 12 weeks
  Regular Pill Counts
Response to iron repletion | 12 weeks
  Hematocrit
Response to iron repletion | 12 weeks
  Iron storage
Response to iron repletion | 12 weeks
  Iron saturation
Response to iron repletion | 12 weeks
  Ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Ala Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon

REFERENCES:
- [Background] Gasche C, Lomer MC, Cavill I, Weiss G. Iron, anaemia, and inflammatory bowel diseases. Gut. 2004 Aug;53(8):1190-7. doi: 10.1136/gut.2003.035758. PMID 15247190
- [Background] Carrier J, Aghdassi E, Cullen J, Allard JP. Iron supplementation increases disease activity and vitamin E ameliorates the effect in rats with dextran sulfate sodium-induced colitis. J Nutr. 2002 Oct;132(10):3146-50. doi: 10.1093/jn/131.10.3146. PMID 12368409
- [Background] Seril DN, Liao J, Yang GY, Yang CS. Oxidative stress and ulcerative colitis-associated carcinogenesis: studies in humans and animal models. Carcinogenesis. 2003 Mar;24(3):353-62. doi: 10.1093/carcin/24.3.353. PMID 12663492
- [Background] Lugg S, Beal F, Nightingale P, Bhala N, Iqbal T. Iron treatment and inflammatory bowel disease: what happens in real practice? J Crohns Colitis. 2014 Aug;8(8):876-80. doi: 10.1016/j.crohns.2014.01.011. Epub 2014 Jan 31. PMID 24486177